CLINICAL TRIAL: NCT03307694
Title: Multi-Angle Compound Shear Wave Elasticity Imaging for the Characterization of Thyroid Nodules
Brief Title: Thyroid Ultrasound Elasticity (TrUE) Imaging
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Stanislav Emelianov, Adjunct Professor, Emory University
Other Study IDs: IRB00092785
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Cancer, Thyroid
Keywords: Cancer; Thyroid nodule; Imaging; Radiology
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasms; Thyroid Nodule | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- MAC-SWEI, standard SWEI, ultrasound: Participants in this group will receive all three imaging techniques
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Shear wave elasticity imaging; Diagnostic Test: Multi-angle compound shear wave elasticity imaging
- Standard SWEI, ultrasound: Participants in this group will receive two imaging techniques
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Shear wave elasticity imaging

INTERVENTIONS:
Diagnostic Test: Ultrasound — All ultrasound images will be acquired by an in-house ultrasound technologist using a Verasonics Vantage (Verasonics Inc., Kirkland, Washington, USA) ultrasound system. During imaging, the technologist will position the Verasonics transducer, under b-mode guidance, in planes overlying the thyroid nodules approximating those obtained during previous clinical ultrasound scans.
Diagnostic Test: Shear wave elasticity imaging — Shear wave elasticity imaging (SWEI) is obtained during the standard ultrasound session. The generation of shear wave images consists of two important steps called "pushing" and "tracking". First, in the "pushing" mode, a long focused ultrasound beam is transmitted to perturb tissue, generating ultrasonic shear waves in tissue that propagate perpendicular to the direction of pushing. In the "tracking" mode, shear wave propagation is observed and recorded. Because the speed of shear waves is a function of Young's modulus, these data reveal information about the stiffness of underlying biological tissue.
  Other Names: SWEI
Diagnostic Test: Multi-angle compound shear wave elasticity imaging — The multi-angle compound SWEI (MAC-SWEI) algorithm, which generates shear images based on multiple angled push beams, has the potential to generate more accurate shear wave images in the context of thyroid imaging. To assess the MAC-SWEI technique, shear wave images will be used to generate estimates of the relative stiffness of lesions via their normalized Young's modulus.
  Other Names: MAC-SWEI
  Groups: MAC-SWEI, standard SWEI, ultrasound

SUMMARY:
In this study the researchers will scan the thyroid nodules of patients scheduled for surgical removal of these nodules. During their preadmission testing, but prior to their surgery, the researchers will perform standard ultrasound and shear wave elasticity imaging (SWEI) scans of the thyroid nodules in these patients. Both images can be generated by the same ultrasound scanner and within the same imaging session without having to switch out any equipment. The results of the SWEI scans will be compared to the definitive diagnosis from pathology obtained after pathologists have examined the removed nodules post-operatively.

DETAILED DESCRIPTION:
Thyroid ultrasound is a first-line procedure to assess patients with thyroid nodules. Unfortunately, standard ultrasound has low sensitivity, and thus low positive predictive value, for malignancy and many patients with thyroid nodules are referred for additional imaging studies or biopsy. Shear wave elasticity imaging (SWEI) is a non-invasive ultrasound technology that allows clinicians to assess the stiffness of tissues. In many solid tumors, increased stiffness is highly specific for underlying malignancy, and preliminary studies have shown this to be true for thyroid malignancies. Both standard sonography and SWEI can be performed on the same ultrasound equipment and within the same imaging session. Therefore, integrating SWEI into standard thyroid diagnostic workflow is a logical approach towards improving the positive predictive value of these first-line sonographic studies. Other studies have demonstrated the ability of SWEI techniques to differentiate benign from malignant thyroid nodules. However, shear wave techniques still need to overcome challenges before they can be successfully integrated into the clinical paradigm. These techniques still struggle to accurately classify follicular carcinomas and few have been validated in patients with multiple thyroid lesions, a scenario which is clinically common. The researchers believe that a multi-angle compound SWEI (MAC-SWEI) algorithm, which generates shear images based on multiple angled push beams, has the potential to generate more accurate shear wave images in the context of thyroid imaging. To this end, this study will perform proof-of-concept studies of MAC-SWEI in thyroid patients undergoing standard ultrasound scans and compare the results of shear wave images to results from corresponding pathology.

Study participants will undergo a single SWEI session within their normally-scheduled preadmission testing during which both standard b-mode and shear images of the thyroid nodule(s) will be acquired. The 36 patients will be randomized to receive MAC-SWEI, standard SWEI, and ultrasound, or only standard SWEI and ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Scheduled to undergo a thyroid biopsy, thyroidectomy, or cervical node biopsy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from patients of the Emory Healthcare system who are scheduled to have a thyroid biopsy, thyroidectomy, or cervical node biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Determination of Malignancy by SWEI Imaging | Pre-operative visit (within 24 hours before surgery, on average)
  As part of the pre-operative visit, participants will have imaging of their thyroid nodules. Established SWEI and MAC-SWEI techniques will be performed to identify malignant thyroid tissue.
Determination of Malignancy by Pathological Proof | Post-surgery (within 10 days after surgery, on average)
  Tissue samples obtained during the participant's thyroid biopsy, thyroidectomy, or cervical node biopsy will be submitted to the pathology lab as part of the clinical standard of care. The pathology report will specify whether or not malignant cells were found in the tissue sample.

SECONDARY OUTCOMES:
Accuracy of differentiating benign from malignant lesions between SWEI techniques | Pre-operative visit (within 24 hours before surgery, on average)
  The ability of MAC-SWEI to differentiate benign from malignant lesions will be compared to the ability of standard SWEI to make this differentiation.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Emelianov, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Univeristy Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No